CLINICAL TRIAL: NCT07332507
Title: Phase 1b Study of Teclistamab in Relapsed/Refractory Plasmablastic Lymphoma
Brief Title: Testing the Effect of Teclistamab on Recurrent Plasmablastic Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-09714; NCI-2025-09714 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-155; 10727 (Other: City of Hope Comprehensive Cancer Center LAO); 10727 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2026-01-09; First posted 2026-01-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Plasmablastic Lymphoma; Refractory Plasmablastic Lymphoma
MeSH Terms: conditions — Plasmablastic Lymphoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (teclistamab) (Experimental): Patients receive teclistamab SC on days 1, 4, and 7 of cycle 1 and on day 1 of remaining cycles. Based on dose level, cycles repeat weekly, every 2 weeks or every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who have achieved a CR by cycle 13 may discontinue study treatment. Patients achieving less than a CR but benefiting from treatment may continue to receive teclistamab beyond 13 cycles in the absence of disease progression, unacceptable toxicity, or achieving a CR. Additionally, patients undergo optional buccal swab collection at baseline and optional blood sample collection throughout the study. Patients also undergo PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Drug: Teclistamab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo buccal swab and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Teclistamab — Given SC
  Other Names: JNJ 64007957; JNJ-64007957; JNJ64007957; Teclistamab-cqyv; Tecvayli

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose, as well as the effectiveness of teclistamab in treating patients with plasmablastic lymphoma that has come back after a period of improvement (recurrent) or that has not responded to previous treatment (refractory). Teclistamab is a bispecific antibody that can bind to two different antigens at the same time. Teclistamab binds to B-cell maturation antigen (BCMA), a protein found on some B-cells and myeloma cells, and CD3 on T-cells (a type of white blood cell) and may interfere with the ability of cancer cells to grow and spread. Giving teclistamab may be safe, tolerable, and/or more effective than usual treatment with radiation or chemotherapy in treating patients with recurrent or refractory plasmablastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximal tolerated dose (MTD) of teclistamab in relapsed/refractory (R/R) plasmablastic lymphoma (PBL).

SECONDARY OBJECTIVES:

I. To estimate the overall response rate (ORR), complete response (CR) rate, progression-free survival (PFS), and overall survival (OS) of teclistamab in R/R PBL.

II. To observe and record anti-tumor activity.

EXPLORATORY OBJECTIVES:

I. To evaluate the utility of B-cell maturation antigen (BCMA) as a biomarker of response to teclistamab in PBL.

II. To evaluate minimum residual disease (MRD) dynamics during treatment.

OUTLINE:

Patients receive teclistamab subcutaneously (SC) on days 1, 4, and 7 of cycle 1 and on day 1 of remaining cycles. Based on dose level, cycles repeat weekly, every 2 weeks or every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who have achieved a complete response (CR) by cycle 13 may discontinue study treatment. Patients achieving less than a CR but benefiting from treatment may continue to receive teclistamab beyond 13 cycles in the absence of disease progression, unacceptable toxicity, or achieving a CR. Additionally, patients undergo optional buccal swab collection at baseline and optional blood sample collection throughout the study. Patients also undergo positron emission tomography (PET)/computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed R/R PBL
* Patients must have measurable disease, defined as at least one bi-dimensionally measurable nodal lesion, defined as ≥ 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extranodal lesion, defined as ≥ 1.0 cm in its longest dimension
* Patients should have ≥ 1 line of prior therapy. This includes at least 1 prior line of chemotherapy or radiation
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of teclistamab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 75,000/mcL
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with central nervous system (CNS) lymphoma are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Based on the mechanism of action, teclistamab may cause fetal harm when administered to a pregnant woman. Females of child-bearing potential (FCBP) should use effective contraception during treatment with teclistamab and for 6 months after the last dose. FCBP should not breast feed during treatment with teclistamab and for 6 months after the last dose. Should a FCBP become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Male patients with a partner who is a FCBP should use effective contraception during treatment and for 3 months after the last dose of teclistamab. Women of childbearing age should not donate eggs and men should not donate sperm for the duration of study participation. Women should not donate eggs for 6 months and men should not donate sperm for 3 months after completion of the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Vaccination with live virus vaccines is not recommended for at least 4 weeks prior to the start of treatment, during treatment and at least 4 weeks after treatment

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and peripheral neuropathy
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to teclistamab
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because teclistamab is a bispecific T-cell antibody agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with teclistamab, breastfeeding should be discontinued if the mother is treated with teclistamab. These potential risks may also apply to other agents used in this study
* Pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation
* Corticosteroid use for purposes other than lymphoma symptom control

  * The use of inhaled corticosteroids is permitted
  * The use of mineralocorticoids for management of orthostatic hypotension is permitted
  * The use of physiologic doses of corticosteroids for management of adrenal insufficiency is permitted
  * Participants who require lymphoma symptom control during screening may receive steroids in the following manner:

    * Up to 100 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days after last dose of study treatment
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. and American Society for Transplantation and Cellular Therapy/Immune Effector Cell Associated Neurotoxicity Syndrome criteria/grading. Descriptive statistics will be employed in the analysis of all safety observations in this study.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years after last dose of study treatment
  Will be assessed by the 2014 Lugano Response Criteria (Cheson et al., 2014). An alternative hypothesis of 40% ORR versus a null hypothesis of 10% will be tested in the dose-expansion cohort. A Simon's Two-Stage Minimax design (Simon, 1989) will be applied to test the hypothesis.
Complete response rate | Up to 2 years after last dose of study treatment
  Will be assessed by the 2014 Lugano Response Criteria (Cheson et al., 2014).
Progression-free survival (PFS) | From start of protocol treatment to time of progressive disease/relapse or death due to any cause, whichever occurs earlier, assessed up to 2 years
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. 95% confidence intervals will be constructed based on log-log transformation.
Overall survival (OS) | From start of protocol treatment to time of death due to any cause, assessed up to 2 years
  OS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. 95% confidence intervals will be constructed based on log-log transformation.

OTHER OUTCOMES:
Utility of B-cell maturation antigen (BCMA) as a biomarker of response | Up to 2 years after last dose of study treatment
  Archival pre-treatment formalin fixed and paraffin embedded tumor samples will be stained with a BCMA immunohistochemistry (IHC) antibody (clone E6D7B) and an H-score will be determined by an expert hematopathologist. Associations between BCMA IHC H-score and response to teclistamab will be determined using a Fisher's exact test at an H-score cutoff of 100.
Impact of minimum residual disease (MRD) on PFS | Up to 2 years after last dose of study treatment
  Impact will be determined by a cycle 3 circulating tumor deoxyribonucleic acid level on 2-year PFS. The Kaplan-Meier method will be used to estimate PFS and a log-rank test will be used to compare the PFS between MRD-positive and MRD-negative groups.

CONTACTS AND LOCATIONS:
Overall Officials: James Godfrey, Principal Investigator — City of Hope Comprehensive Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm